CLINICAL TRIAL: NCT06318182
Title: The Effect of Training Based on the Health Belief Model on Testicular Self-Examination Awareness and Health Beliefs in Young Men
Brief Title: Testicular Self-Examination Awareness in Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Emre Keles, Research Assistant, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NCT-SBF-EK-001
Record Dates: First submitted 2024-02-19; First posted 2024-03-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-03

CONDITIONS: Testicular Cancer
Keywords: awareness; health behavior; testicular cancer
MeSH Terms: conditions — Testicular Neoplasms; Health Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training group (Experimental): Group receiving training based on SIMTEKEP program
  Interventions: Other: Education
- Control group (No Intervention): The group that did not receive training based on the SIMTEKEP program

INTERVENTIONS:
Other: Education — Young men who are included in the research sample and agree to participate in the study will be given training within the scope of the health belief model.
  Arms: Training group

SUMMARY:
This study aims to determine the effect of education based on the health belief model on testicular self-examination awareness and health beliefs in young men.

H0 Hypothesis: Education based on the health belief model has no effect on the awareness of testicular self-examination and health beliefs about testicular self-examination of young men in the experimental and control groups.

H1a Hypothesis: The training based on the health belief model will increase the awareness of young men in the experimental group about testicular self-examination compared to those in the control group.

H1b Hypothesis: The training based on the health belief model will increase the mean scores of the sensitivity subscale of young men in the experimental group compared to those in the control group.

H1c Hypothesis: The training based on the health belief model will increase the mean scores of the benefit subscale of young men in the experimental group compared to those in the control group.

H1d Hypothesis: The training based on the health belief model will increase the mean scores of the seriousness subscale of young men in the experimental group compared to those in the control group.

H1e Hypothesis: The training based on the health belief model will decrease the mean scores of the barriers subscale of young men in the experimental group compared to those in the control group.

H1f Hypothesis: The training based on the health belief model will increase the mean scores of the health motivation subscale of young men in the experimental group compared to those in the control group.

H1g Hypothesis: The training based on the health belief model will increase the mean scores of the self-efficacy subscale of young men in the experimental group compared to those in the control group.

DETAILED DESCRIPTION:
The research data will be obtained from students of Hitit University Faculty of Health Sciences, Department of Child Development, Department of Health Management, Department of Social Work, and Department of Nutrition and Dietetics between 20 November 2023 and 15 July 2024.

Pre-intervention phase: Data collection forms were applied to n=120 participants who met the inclusion criteria and accepted the study (pretest).Experimental (n=60) and control (n=60) groups were formed by drawing lots among the participants.

"Testicular Cancer Education Program Based on Health Belief Model (SİMTEKEP)," prepared by the researcher based on the literature, was carried out in four sessions. In the first session (45-60 minutes), "Male reproductive organs, testicular cancer and its symptoms (PERCEPTION OF SENSITIVITY)"; in the second session (45-60 minutes), "Treatment of testicular cancer and its negative effects (PERCEPTION OF SERIOUSNESS)"; in the third session (45-60 minutes) "Early diagnosis and Testicular Self-Examination (PERCEPTION OF BENEFIT and SELF-EFFICIENCY)"; and in the last session (45-60 minutes), "Testicular Self-Examination (PERCEPTION OF OBSTACLE)" topics were discussed. After the training, reminder messages were sent to the participants once a week.

Post-intervention phase: At the end of the third month after the intervention, data collection forms will be applied again, and the research process will be completed (Monitoring).

ELIGIBILITY:
Inclusion Criteria:

* Being male
* Being between the ages of 18 and 35
* Studying at Hitit University Faculty of Health Sciences
* Not having attended a course or training program on testicular cancer.

Exclusion Criteria:

* Being under 18 years of age or over 35 years of age
* Being a student in the Department of Nursing
* Participating in a course or training program on testicular cancer
* Having testicular cancer

Ages: 15 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Since the subject is related to testicular cancer and should be evaluated from the perspective of men, only men were included in the study.
Enrollment: 120 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Demographic information and testicular cancer questionnaire | one week
  As a pre-test, a survey form consisting of 21 questions prepared by the researcher by scanning the literature.
Testicular Cancer Knowledge Test | one week
  As a pre-test, a knowledge test consisting of 20 questions prepared by the researcher by scanning the literature.
  There are true and false statements in the Testicular Cancer Knowledge Test. Participants are asked to evaluate these statements as true or false. Each correct answer is evaluated as 1 point, and an incorrect answer is evaluated as 0 points.
Health Beliefs Scale for Testicular Cancer and Testicular Self-Examination | one week
  As a pre-test, Health Beliefs Scale for Testicular Cancer and Testicular Self-Examination
  The minimum score from the scale is 37 and the maximum is 185. Each dimension of the scale is evaluated separately, and as the score increases, positive behavior increases.

SECONDARY OUTCOMES:
For the control group, Testicular Cancer Knowledge Test | three months
  The Testicular Cancer Knowledge Test was administered as a posttest.
For the control group, Health Beliefs Scale for Testicular Cancer and Testicular Self-Examination | three months
  The Health Beliefs Scale for Testicular Cancer and Testicular Self-Examination was administered as a posttest.

OTHER OUTCOMES:
Testicular Cancer Knowledge Test | three months
  The Testicular Cancer Knowledge Test will be administered as a follow-up test.
Health Beliefs Scale for Testicular Cancer and Testicular Self-Examination | three months
  The Health Beliefs Scale for Testicular Cancer and Testicular Self-Examination will be administered as a follow-up test.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Keles, Principal Investigator — Hitit University; Birsen Altay, Study Director — Ondokuz Mayıs University
Locations (1):
- Hitit University, Çorum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Informed Consent Form (ICF) information will be shared.